CLINICAL TRIAL: NCT02441829
Title: A Phase 1 Open-Label, Parallel-Group, Adaptive, Single Dose Study to Evaluate the Pharmacokinetics of GS-6615 in Subjects With Normal and Impaired Renal Function
Brief Title: Pharmacokinetics of Eleclazine in Adults With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-372-1589; 2014-005267-32 (EudraCT Number)
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Long QT Syndrome
Keywords: Renal Impairment
MeSH Terms: conditions — Long QT Syndrome; Renal Insufficiency | interventions — eleclazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild Renal Impairment (CLcr 60-89 mL/min) (Experimental): Participants with mild renal impairment and matched control participants with normal renal function will receive a single dose of eleclazine 30 mg (5 x 6 mg tablets).
  Interventions: Drug: Eleclazine
- Moderate Renal Impairment (CLcr 30-59 mL/min) (Experimental): Participants with moderate impairment and matched control participants with normal renal function will receive a single dose of eleclazine 30 mg (5 x 6 mg tablets).
  Interventions: Drug: Eleclazine
- Severe Renal Impairment (CLcr 15-29 mL/min) (Experimental): Participants with severe renal impairment and matched control participants with normal renal function will receive a single dose of eleclazine 30 mg (5 x 6 mg tablets).
  Interventions: Drug: Eleclazine

INTERVENTIONS:
Drug: Eleclazine — Eleclazine tablets administered orally in morning with food
  Other Names: GS-6615

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, and tolerability of a single oral dose of eleclazine and its metabolite, GS-623134, in participants with normal and impaired renal function. Participants in the healthy control group will be matched to participants with impaired renal function by age (± 5 years), gender, and body mass index (± 10%).

ELIGIBILITY:
Inclusion Criteria:

All Individuals:

* Be a nonsmoker or consume < 20 cigarettes per day
* Have a calculated body mass index (BMI) from 18 to 36 kg/m^2, inclusive, at study screening
* Have either a normal 12-lead electrocardiogram (ECG) or one with abnormalities that are considered clinically insignificant by the investigator
* Screening labs within defined thresholds

Individuals with mild, moderate, or severe renal impairment must also meet the following additional inclusion criteria to be eligible for participation in this study:

* Must have diagnosis of chronic (> 6 months), stable renal impairment with no clinically significant changes within 3 months (90 days) prior to study drug administration (Day 1)
* Individuals with severe renal impairment, creatinine clearance (CLcr) must be 15-29 mL/min, inclusive (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at the screening evaluation. If an individual's score changes during the course of the study, the score at screening will be used for classification.
* Individuals with moderate renal impairment, CLcr must be 30-59 mL/min, inclusive (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at the screening evaluation. If an individual's score changes during the course of the study, the score at screening will be used for classification.
* Individuals with mild renal impairment , CLcr must be 60-89, inclusive mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at the screening evaluation. If an individual's score changes during the course of the study, the score at screening will be used for classification.

Individuals with normal renal function must also meet the following additional inclusion criteria to be eligible for participation in this study:

* Must, in the opinion of the Investigator, be in good health based upon medical history, physical examination, vital signs, and screening laboratory evaluations
* Must have an CLcr of ≥ 90 mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at the screening evaluation.

Exclusion Criteria:

* History of meningitis or encephalitis, epilepsy, seizures, migraines, tremors, myoclonic jerks, narcolepsy, obstructive sleep apnea, anxiety, syncope, head injuries or a family history of seizures
* Presence or history of cardiovascular disease (including history of myocardial infarction based on ECG and/or clinical history, any history of ventricular tachycardia, congestive heart failure, cardiomyopathy, or left ventricular ejection fraction < 40%), cardiac conduction abnormalities, a family history of Long QT Syndrome, or unexplained death in an otherwise healthy individual between the ages of 1 and 30 years
* Syncope, palpitations, or unexplained dizziness
* Implanted defibrillator or pacemaker
* Medical history of renal carcinoma or hepatorenal syndrome.
* Individuals receiving or anticipating use of hemodialysis, peritoneal dialysis, or any other renal replacement therapy or other medical procedure that serves as a surrogate for renal function during the study.
* Individuals with fluctuating or rapidly deteriorating renal function. Assessment of the stability of the individual's renal function will be determined by the investigator.
* Renal allograft recipients
* Experienced hypertensive crisis, required the addition of ≥1 antihypertensive drug, or required more intensive antihypertensive therapy (eg, addition of a new drug class) in the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics (PK) profiles of eleclazine and its metabolite GS-623134: AUC_0-inf and Cmax | Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, 14, 24, 36, 48, 72, 96, 120 hours, 15, 29, 43, and 57 days postdose on Day 1
  This endpoint will measure the plasma PK profiles of eleclazine and GS-623134. PK parameters that will be measured include AUC_0-inf and Cmax.

SECONDARY OUTCOMES:
Safety profile of eleclazine as measured by incidence of adverse events and laboratory abnormalities | Up to 58 days

CONTACTS AND LOCATIONS:
Overall Officials: Brian McNabb, MD, Study Director — Gilead Sciences
Locations (7):
- United States (5):
  - DeLand, Florida
  - Miami, Florida
  - Orlando, Florida
  - Saint Paul, Minnesota
  - Kansas City, Missouri
- Chisinau, Moldova
- Bucharest, Romania